CLINICAL TRIAL: NCT03837743
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Proof of Concept Comparison Study of the Safety and Efficacy of DUR-928 Topical Solution With Occlusion in Subjects With Mild to Moderate Plaque Psoriasis
Brief Title: Safety and Efficacy Study of DUR-928 Topical Solution in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C928-015
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Results first posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DUR-928 Topical Solution (Experimental): DUR-928 Topical Solution applied topically once daily to one target lesion on an arm for approximately four weeks.
  Interventions: Drug: DUR-928 Topical Solution
- Vehicle Topical Solution (Placebo Comparator): Vehicle Topical Solution applied topically once daily to one target lesion on an arm for approximately four weeks.
  Interventions: Drug: Vehicle Topical Solution

INTERVENTIONS:
Drug: DUR-928 Topical Solution — Topical solution containing active drug
  Arms: DUR-928 Topical Solution
Drug: Vehicle Topical Solution — Topical solution containing no active drug
  Arms: Vehicle Topical Solution

SUMMARY:
This Phase 2 study has been designed to determine and compare the safety, tolerability, and efficacy of DUR-928 topical solution with that of the vehicle topical solution when applied once daily for approximately four weeks in subjects with plaque psoriasis. Subjects will be instructed (randomly assigned) to apply DUR-928 solution to a target lesion on one arm and vehicle solution to a target lesion on the opposite arm once daily for up to four weeks. Subjects will occlude the treated areas for approximately two hours after each application.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or non-pregnant female 18 years of age or older.
2. Subject has provided written informed consent.
3. Subject has a clinical diagnosis of stable mild to moderate plaque psoriasis for at least two months.
4. Females must be post-menopausal, surgically sterile, or use an effective method of birth control. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 2/Baseline.
5. Males (or their female partner) must agree to use an effective method of birth control throughout the study.
6. Subject has two similar contralateral Target Plaques.
7. Subject is willing and able to apply the test article(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
8. Subject, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation of the plaque psoriasis or exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
3. Subject has guttate, pustular, erythrodermic, inverse, or other non-plaque forms of psoriasis.
4. Subject has psoriasis beyond the two Target Plaques that, in the investigator's opinion, could not be reasonably managed with only a bland emollient during the study.
5. Subject is currently enrolled in an investigational drug or device study.
6. Subject has been previously enrolled in this study and treated with test article.

Other protocol-defined inclusion and exclusion criteria assessed by the study staff may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Andrasfay, Study Director — Therapeutics, Inc.
Locations (5):
- United States (5):
  - Site 01, San Diego, California
  - Site 04, Miami, Florida
  - Site 05, Tampa, Florida
  - Site 02, Plainfield, Indiana
  - Site 03, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-site study conducted at five sites in the United States of America. Date first subject enrolled: March 20, 2019 and date last subject completed: November 7, 2019.
Units Other Than Participants: lesions
Groups:
- DUR-928 Topical Solution and Vehicle Topical Solution: DUR-928 Topical Solution and Vehicle Topical Solution separately applied topically once daily to one target lesion on an arm of a subject for approximately four weeks. Each arm of a subject containing one target lesion was allocated to a different intervention.
  DUR-928 Topical Solution: Topical solution containing active drug
  Vehicle Topical Solution: Topical solution containing no active drug
Period: Overall Study
Arm/Group | DUR-928 Topical Solution and Vehicle Topical Solution
Started | 25; 50 lesions
DUR-928 Topical Solution Lesion | 25; 25 lesions
Vehicle Topical Solution Lesion | 25; 25 lesions
Completed | 22; 44 lesions
Not Completed | 3; 6 lesions
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- DUR-928 Topical Solution and Vehicle Topical Solution: DUR-928 Topical Solution and Vehicle Topical Solution applied topically once daily to one target lesion on an arm for approximately four weeks.
  DUR-928 Topical Solution: Topical solution containing active drug Vehicle Topical Solution: Topical solution containing no active drug
Arm/Group | DUR-928 Topical Solution and Vehicle Topical Solution
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline as Assessed on the Investigator's Global Assessment (IGA) Score.
Description: The IGA of the Target Plaques will be determined on a 5-point scale. 0=Clear; 1=Almost Clear; 2=Mild; 3=Moderate; 4=Severe
Time Frame: Up to Day 57 (assessed at Baseline, and Weeks 1,2,3,4,5,7,8, change from baseline to week 4 and 8 reported)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DUR-928 Topical Solution | Vehicle Topical Solution
Number analyzed (Participants) | 25 | 25
score on a scale
  Week 4 (change from baseline) | -0.8 (0.83) | -1.0 (0.93)
  Week 8 (change from baseline) | -0.6 (1.00) | -0.8 (1.10)
Statistical Analysis 1: Comparison: DUR-928 Topical Solution vs Vehicle Topical Solution; Difference in Change (week 4); Test type: Superiority; p = 0.022, Paired t-test; Mean Difference (Final Values) = 0.2, Standard Deviation 0.42
Statistical Analysis 2: Comparison: DUR-928 Topical Solution vs Vehicle Topical Solution; Difference in Change (week 8); Test type: Superiority; p = 0.296, Paired t-test; Mean Difference (Final Values) = 0.2, Standard Deviation 0.80

2. Secondary Outcome: The Change From Baseline as Assessed on the Clinical Signs of Psoriasis (Plaque Elevation, Scaling, and Erythema)
Description: Each clinical sign (plaque elevation, scaling, erythema) will be graded on a 5-point scale.0=Clear; 1=Almost Clear; 2=Mild; 3=Moderate; 4=Severe.
Time Frame: Up to Day 57 (assessed at Baseline, and Weeks 1,2,3,4,5,7,8, change from baseline to week 4 and 8 reported)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DUR-928 Topical Solution | Vehicle Topical Solution
Number analyzed (Participants) | 25 | 25
score on a scale
  Week 4 (Clinical Signs of Psoriasis - Plaque Elevation-Change from Baseline) | -1.0 (0.88) | -1.2 (0.94)
  Week 8 (Clinical Signs of Psoriasis - Plaque Elevation-Change from Baseline) | -0.7 (0.98) | -0.9 (1.06)
  Week 4 (Clinical Signs of Psoriasis - scaling-Change from Baseline) | -0.8 (0.89) | -1.1 (1.06)
  Week 8 (Clinical Signs of Psoriasis - scaling-Change from Baseline) | -0.6 (0.95) | -0.8 (1.18)
  Week 4 (Clinical Signs of Psoriasis - erythema-Change from Baseline) | -1.0 (0.88) | -1.1 (1.00)
  Week 8 (Clinical Signs of Psoriasis - erythema-Change from Baseline) | -0.9 (0.97) | -1.1 (0.97)

3. Secondary Outcome: The Change From Baseline as Assessed on the Local Psoriasis Severity Index (LPSI)
Description: The LPSI is a sum of all three parameters (sum range of 0-12, with 12 being a worse outcome). Three parameters are plaque elevation, scaling, and erythema, each rated 0-4, 0=clear to 4=severe.
Time Frame: Up to Day 57 (assessed at Baseline, and Weeks 1,2,3,4,5,7,8, change from baseline to week 4 and 8 reported)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DUR-928 Topical Solution | Vehicle Topical Solution
Number analyzed (Participants) | 25 | 25
score on a scale
  week 4 (change from Baseline) | -2.7 (2.40) | -3.4 (2.76)
  week 8 (change from Baseline) | -2.3 (2.69) | -2.8 (3.05)

4. Secondary Outcome: The Change From Baseline as Assessed by the Target Plaque Area.
Description: The surface areas of Target Plaque A (plaque on left arm) and Target Plaque B (plaque on right arm) will be measured.
Time Frame: Up to Day 57 (assessed at Baseline, and Weeks 2,4,8, change from baseline to week 4 and 8 reported)
Population: ITT population
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | DUR-928 Topical Solution | Vehicle Topical Solution
Number analyzed (Participants) | 25 | 25
cm^2
  Week 4 (change from Baseline) | -2.5 (11.02) | -7.4 (10.88)
  Week 8 (change from Baseline) | -5.8 (10.26) | -8.3 (7.85)

5. Secondary Outcome: The Change From Baseline as Assessed on the Itch Numeric Rating Scale (I-NRS) for Pruritus.
Description: The I-NRS score is based on an 11-point scale where 0 represents "no itching" and 10 represents "worst itch imaginable."
Time Frame: Up to Day 57 (assessed at Baseline, and Weeks 2,4,8, change from baseline to week 4 and 8 reported)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DUR-928 Topical Solution | Vehicle Topical Solution
Number analyzed (Participants) | 25 | 25
units on a scale
  Week 4 (change from baseline) | -1.7 (2.19) | -1.7 (1.84)
  Week 8 (change from baseline) | -1.6 (2.34) | -1.5 (2.11)

6. Other Pre Specified Outcome: The Change From Baseline as Assessed on the Target Plaque Comparison
Description: The Target Plaque Comparison is scored on a 3-point scale: 1A = Target Plaque A is better than Target Plaque B, 0 = Target Plaque A is the same as Target Plaque B, and 1B = Target Plaque A is worse than Target Plaque B.
Time Frame: Up to Day 57 (assessed at Baseline, and Weeks 1,2,3,4,5,7,8, change from baseline to week 4 and 8 reported)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | DUR-928 Topical Solution and Vehicle Topical Solution
Number analyzed (Participants) | 23
participants
  Week 4 : Active Better | 2
  Week 4 : Same | 13
  Week 4 : Active Worse | 8
  Week 8 : Active Better: number analyzed (Participants) | 22
  Week 8 : Active Better | 3
  Week 8 : Same: number analyzed (Participants) | 22
  Week 8 : Same | 11
  Week 8 : Active Worse: number analyzed (Participants) | 22
  Week 8 : Active Worse | 8

ADVERSE EVENTS:
Time Frame: Up to Day 57
Description: Treatment emergent adverse events (TEAE) were collected for all subjects. Information on the treatment arm was only collected if the TEAE was local to the application site.
Groups:
- DUR-928 Topical Solution and Vehicle Topical Solution, Safety Population: DUR-928 Topical Solution and Vehicle Topical Solution applied topically once daily to one target lesion on an arm for approximately four weeks. This group reflects all TEAEs collected for the safety population, including those that are treatment application site specific.
- DUR-928 Topical Solution, Safety Population Experiencing a TEAE at the Treatment Application Site.: DUR-928 Topical Solution: Topical solution containing active drug applied topically once daily to one target lesion on an arm for approximately four weeks.
  This treatment arm was only reported if the TEAE was local to the treatment application site.
- Vehicle Topical Solution, Safety Population Experiencing a TEAE at the Treatment Application Site.: Vehicle Topical Solution: Topical solution containing no active drug applied topically once daily to one target lesion on an arm for approximately four weeks.
  This treatment arm was only reported if the TEAE was local to the treatment application site.
Arm/Group | DUR-928 Topical Solution and Vehicle Topical Solution, Safety Population | DUR-928 Topical Solution, Safety Population Experiencing a TEAE at the Treatment Application Site. | Vehicle Topical Solution, Safety Population Experiencing a TEAE at the Treatment Application Site.
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 11/25 | 4/25 | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | DUR-928 Topical Solution and Vehicle Topical Solution, Safety Population (N=25) | DUR-928 Topical Solution, Safety Population Experiencing a TEAE at the Treatment Application Site. (N=25) | Vehicle Topical Solution, Safety Population Experiencing a TEAE at the Treatment Application Site. (N=25)
Diarrhoea (Gastrointestinal disorders) | 1 | 0/0 | 0/0
Application site erythema (General disorders) | 1 | 1 | 1
Application site fissure (General disorders) | 1 | 1 | 1
Application site haemorrhage (General disorders) | 1 | 1 | 1
Application site injury (General disorders) | 1 | 1 | 0
Application site pain (General disorders) | 1 | 1 | 1
Application site pruritus (General disorders) | 1 | 1 | 1
Ear infection (Infections and infestations) | 1 | 0/0 | 0/0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0/0 | 0/0
Blood urine (Investigations) | 1 | 0/0 | 0/0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0/0 | 0/0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0/0 | 0/0
Headache (Nervous system disorders) | 1 | 0/0 | 0/0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0/0 | 0/0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0/0 | 0/0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0/0 | 0/0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0/0 | 0/0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0/0 | 0/0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0/0 | 0/0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure agreement provides that if sponsor has not submitted a manuscript for publication within 12 months after the date of data lock and analysis at study completion at all sites, the PI can review results communications prior to public release and can embargo communications regarding trial results for a period up to 120 days from the time submitted to the sponsor for review. The PI cannot disclose SPONSOR Confidential Information without prior consent.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03837743/Prot_SAP_000.pdf